CLINICAL TRIAL: NCT03451474
Title: Restoring Hand Function Utilizing Nerve Transfers in Persons With Cervical Spinal Cord Injuries
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-17-0081
Record Dates: First submitted 2018-02-08; First posted 2018-03-01 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Cervical Spinal Cord Injury; Spinal Cord Injuries; Traumatic Spinal Cord Compression
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Upper extremity nerve transfer surgery (Experimental): Upper extremity nerve transfer surgery is a surgical procedure where axons from an intact, functioning upper extremity peripheral nerve are moved to a target muscle that demonstrates significant weakness or paralysis as a result of spinal cord injury. After allowing time for recovery from surgery and for nerve growth to occur, the patient undergoes hand/occupational therapy in order to retrain motor skills.
  Interventions: Procedure: Upper extremity nerve transfer surgery

INTERVENTIONS:
Procedure: Upper extremity nerve transfer surgery — Upper extremity nerve transfer surgery is a surgical procedure where axons from an intact, functioning upper extremity peripheral nerve are moved to a target muscle that demonstrates significant weakness or paralysis as a result of spinal cord injury. After allowing time for recovery from surgery and for nerve growth to occur, the patient undergoes hand/occupational therapy in order to retrain motor skills.

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of nerve transfer surgery for restoring hand function as a therapy for patients with cervical spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* American Spinal Injury Association (ASIA) grade of A, B, or C, or with a diagnosis of central cord syndrome, showing minimal to no evidence of functional improvement in motor examination after at least 6 months of non-operative therapy post-injury
* >6 months post-injury
* International Classification of Surgery of the Hand in Tetraplegia (ICSHT) category 0-4
* Cervical spinal cord injury resulting in arm & hand functional impairment, with at least preserved elbow flexion
* Physically and mentally willing and able to comply with study protocol
* Lives in the immediate area and has no plans to relocate
* Provides informed consent and HIPAA release of medical information

Exclusion Criteria:

* Active infection
* Any return or ongoing clinical recovery of distal motor function within 6 months after injury
* Physically/mentally compromised
* Systemic disease that would affect the patient's welfare or the research study
* Immunologically suppressed or immunocompromised
* Currently undergoing long-term steroid therapy
* Active malignancy
* Pending litigation or receiving Workers Compensation related to injury or accident
* Pregnancy
* Significant contractures and/or limitations in passive range of motion in the arm or hand
* Poorly controlled upper extremity spasticity
* Uncontrolled pain or hypersensitivity
* Previous or current injury preventing use of tendon transfers to restore upper extremity function
* History of brachial plexus injury or systemic neuropathic process
* In the opinion of the Principal Investigator the subject would not be a candidate for the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Upper extremity muscle strength of right arm as assessed by the Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) strength subscale | Pre-operative
  The GRASSP is a measure of upper extremity strength, sensation, and grip that is specific to patients with tetraplegia. It consists of 5 subscales for each upper extremity, and this measure will report the strength subscale (manual muscle testing of 10 muscles in right arm - subscale total score encompasses all 10 muscles). The strength subscale total score ranges from 0 to 50. The GRASSP will be administered by the nurses or physical therapist involved in the study.
Upper extremity muscle strength of right arm as assessed by the Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) strength subscale | post-operative at 2 weeks
  The GRASSP is a measure of upper extremity strength, sensation, and grip that is specific to patients with tetraplegia. It consists of 5 subscales for each upper extremity, and this measure will report the strength subscale (manual muscle testing of 10 muscles in right arm - subscale total score encompasses all 10 muscles). The strength subscale total score ranges from 0 to 50. The GRASSP will be administered by the nurses or physical therapist involved in the study.
Upper extremity muscle strength of right arm as assessed by the Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) strength subscale | post-operative at 3 months
  The GRASSP is a measure of upper extremity strength, sensation, and grip that is specific to patients with tetraplegia. It consists of 5 subscales for each upper extremity, and this measure will report the strength subscale (manual muscle testing of 10 muscles in right arm - subscale total score encompasses all 10 muscles). The strength subscale total score ranges from 0 to 50. The GRASSP will be administered by the nurses or physical therapist involved in the study.
Upper extremity muscle strength of right arm as assessed by the Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) strength subscale | post-operative at 6 months
  The GRASSP is a measure of upper extremity strength, sensation, and grip that is specific to patients with tetraplegia. It consists of 5 subscales for each upper extremity, and this measure will report the strength subscale (manual muscle testing of 10 muscles in right arm - subscale total score encompasses all 10 muscles). The strength subscale total score ranges from 0 to 50. The GRASSP will be administered by the nurses or physical therapist involved in the study.
Upper extremity muscle strength of right arm as assessed by the Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) strength subscale | post-operative at 12 months
  The GRASSP is a measure of upper extremity strength, sensation, and grip that is specific to patients with tetraplegia. It consists of 5 subscales for each upper extremity, and this measure will report the strength subscale (manual muscle testing of 10 muscles in right arm - subscale total score encompasses all 10 muscles). The strength subscale total score ranges from 0 to 50. The GRASSP will be administered by the nurses or physical therapist involved in the study.
Upper extremity muscle strength of right arm as assessed by the Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) strength subscale | post-operative at 24 months
  e GRASSP is a measure of upper extremity strength, sensation, and grip that is specific to patients with tetraplegia. It consists of 5 subscales for each upper extremity, and this measure will report the strength subscale (manual muscle testing of 10 muscles in right arm - subscale total score encompasses all 10 muscles). The strength subscale total score ranges from 0 to 50. The GRASSP will be administered by the nurses or physical therapist involved in the study.
Upper extremity muscle strength of left arm as assessed by the Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) strength subscale | Pre-operative
  The GRASSP is a measure of upper extremity strength, sensation, and grip that is specific to patients with tetraplegia. It consists of 5 subscales for each upper extremity, and this measure will report the strength subscale (manual muscle testing of 10 muscles in left arm - subscale total score encompasses all 10 muscles). The strength subscale total score ranges from 0 to 50. The GRASSP will be administered by the nurses or physical therapist involved in the study.
Upper extremity muscle strength of left arm as assessed by the Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) strength subscale | post-operative at 2 weeks
  The GRASSP is a measure of upper extremity strength, sensation, and grip that is specific to patients with tetraplegia. It consists of 5 subscales for each upper extremity, and this measure will report the strength subscale (manual muscle testing of 10 muscles in right arm - subscale total score encompasses all 10 muscles). The strength subscale total score ranges from 0 to 50. The GRASSP will be administered by the nurses or physical therapist involved in the study.
Upper extremity muscle strength of left arm as assessed by the Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) strength subscale | post-operative at 3 months
  The GRASSP is a measure of upper extremity strength, sensation, and grip that is specific to patients with tetraplegia. It consists of 5 subscales for each upper extremity, and this measure will report the strength subscale (manual muscle testing of 10 muscles in right arm - subscale total score encompasses all 10 muscles). The strength subscale total score ranges from 0 to 50. The GRASSP will be administered by the nurses or physical therapist involved in the study.
Upper extremity muscle strength of left arm as assessed by the Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) strength subscale | post-operative at 6 months
  The GRASSP is a measure of upper extremity strength, sensation, and grip that is specific to patients with tetraplegia. It consists of 5 subscales for each upper extremity, and this measure will report the strength subscale (manual muscle testing of 10 muscles in right arm - subscale total score encompasses all 10 muscles). The strength subscale total score ranges from 0 to 50. The GRASSP will be administered by the nurses or physical therapist involved in the study.
Upper extremity muscle strength of left arm as assessed by the Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) strength subscale | post-operative at 12 months
  The GRASSP is a measure of upper extremity strength, sensation, and grip that is specific to patients with tetraplegia. It consists of 5 subscales for each upper extremity, and this measure will report the strength subscale (manual muscle testing of 10 muscles in right arm - subscale total score encompasses all 10 muscles). The strength subscale total score ranges from 0 to 50. The GRASSP will be administered by the nurses or physical therapist involved in the study.
Upper extremity muscle strength of left arm as assessed by the Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) strength subscale | post-operative at 24 months
  The GRASSP is a measure of upper extremity strength, sensation, and grip that is specific to patients with tetraplegia. It consists of 5 subscales for each upper extremity, and this measure will report the strength subscale (manual muscle testing of 10 muscles in right arm - subscale total score encompasses all 10 muscles). The strength subscale total score ranges from 0 to 50. The GRASSP will be administered by the nurses or physical therapist involved in the study.

SECONDARY OUTCOMES:
Motor neuron signaling as assessed by electromyography (EMG) | Pre-operative, post-operative at 6 months, 1 year, and 2 years
  Quantitative assessment of motor neuron signalling
Strength as assessed by Manual Muscle Testing (MMT) | Pre-operative (5 repeated measurements over 2 months), post-operative at 2 weeks, 3 months, 6 months, 12 months, and 24 months
  MMT will be assessed by the physicians, nurses, or physical therapist involved in the study.
Strength as assessed by Hand Held Dynamometry (HHD) | Pre-operative (5 repeated measurements over 2 months), post-operative at 2 weeks, 3 months, 6 months, 12 months, and 24 months
  Hand held dynamometry (via a "make test") will be used to assess strength.
Strength as assessed by the American Spinal Injury Association (ASIA) Upper Extremity Motor Score (UEMS) | Pre-operative (5 repeated measurements over 2 months), post-operative at 2 weeks, 3 months, 6 months, 12 months, and 24 months
  The ASIA UEMS is a sum of the motor scores for 5 key upper extremity muscles on both the right and left side (each key muscle is a functionally significant representation of a spinal cord segment). The strength of each key muscle on both the right and left side is graded from 0 to 5, with total scores ranging from 0 to 50.The UEMS will be determined in accordance with the International Standards for Neurological Classification of SCI examination guidelines by the physicians, nurses, or physical therapist.
Dorsal sensation as assessed by the Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) dorsal sensation subscale | Pre-operative (5 repeated measurements over 2 months), post-operative at 2 weeks, 3 months, 6 months, 12 months, and 24 months
  The GRASSP is a measure of upper extremity strength, sensation, and grip that is specific to patients with tetraplegia. It consists of 5 subscales for each upper extremity: strength (manual muscle testing of 10 muscles in right and left arms - subscale total score encompasses all 10 muscles), dorsal sensation, palmar sensation (measured with Semmes-Weinstein monofilaments), qualitative grasp, and quantitative grasp. Total score (which includes all subscale scores) ranges from 0 to 116 for each upper extremity (right or left arm). The dorsal sensation subscale total score ranges from 0 to 12. The GRASSP will be administered by the nurses or physical therapist involved in the study.
Palmar sensation as assessed by the Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) palmar sensation subscale | Pre-operative (5 repeated measurements over 2 months), post-operative at 2 weeks, 3 months, 6 months, 12 months, and 24 months
  The GRASSP is a measure of upper extremity strength, sensation, and grip that is specific to patients with tetraplegia. It consists of 5 subscales for each upper extremity: strength (manual muscle testing of 10 muscles in right and left arms - subscale total score encompasses all 10 muscles), dorsal sensation, palmar sensation (measured with Semmes-Weinstein monofilaments), qualitative grasp, and quantitative grasp. Total score (which includes all subscale scores) ranges from 0 to 116 for each upper extremity (right or left arm). The palmar sensation subscale total score ranges from 0 to 12. The GRASSP will be administered by the nurses or physical therapist involved in the study.
Qualitative grasp as assessed by the Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) qualitative grasp subscale | Pre-operative (5 repeated measurements over 2 months), post-operative at 2 weeks, 3 months, 6 months, 12 months, and 24 months
  The GRASSP is a measure of upper extremity strength, sensation, and grip that is specific to patients with tetraplegia. It consists of 5 subscales for each upper extremity: strength (manual muscle testing of 10 muscles in right and left arms - subscale total score encompasses all 10 muscles), dorsal sensation, palmar sensation (measured with Semmes-Weinstein monofilaments), qualitative grasp, and quantitative grasp. Total score (which includes all subscale scores) ranges from 0 to 116 for each upper extremity (right or left arm). The qualitative grasp subscale total score ranges from 0 to 12. The GRASSP will be administered by the nurses or physical therapist involved in the study.
Quantitative grasp as assessed by the Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) quantitative grasp subscale | Pre-operative (5 repeated measurements over 2 months), post-operative at 2 weeks, 3 months, 6 months, 12 months, and 24 months
  The GRASSP is a measure of upper extremity strength, sensation, and grip that is specific to patients with tetraplegia. It consists of 5 subscales for each upper extremity: strength (manual muscle testing of 10 muscles in right and left arms - subscale total score encompasses all 10 muscles), dorsal sensation, palmar sensation (measured with Semmes-Weinstein monofilaments), qualitative grasp, and quantitative grasp. Total score (which includes all subscale scores) ranges from 0 to 116 for each upper extremity (right or left arm). The quantitative grasp subscale total score ranges from 0 to 30. The GRASSP will be administered by the nurses or physical therapist involved in the study.
Total Score on the Graded Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) scale | Pre-operative (5 repeated measurements over 2 months), post-operative at 2 weeks, 3 months, 6 months, 12 months, and 24 months
  The GRASSP is a measure of upper extremity strength, sensation, and grip that is specific to patients with tetraplegia. It consists of 5 subscales for each upper extremity: strength (manual muscle testing of 10 muscles in right and left arms - subscale total score encompasses all 10 muscles), dorsal sensation, palmar sensation (measured with Semmes-Weinstein monofilaments), qualitative grasp, and quantitative grasp. Total score (which includes all subscale scores) ranges from 0 to 116 for each upper extremity (right or left arm). The GRASSP will be administered by the nurses or physical therapist involved in the study.
Function (self-care) as assessed by the Spinal Cord Independence Measure III Self Report (SCIM III SR) questionnaire | Pre-operative (5 repeated measurements over 2 months), post-operative at 2 weeks, 3 months, 6 months, 12 months, and 24 months
  The SCIM III SR is a measure of independence with activities across 3 subscales: self-care, respiration and sphincter management, and mobility. The self-care subscale ranges from 0 to 20.
Function (respiration and sphincter management) as assessed by the Spinal Cord Independence Measure III Self Report (SCIM III SR) questionnaire | Pre-operative (5 repeated measurements over 2 months), post-operative at 2 weeks, 3 months, 6 months, 12 months, and 24 months
  The SCIM III SR is a measure of independence with activities across 3 subscales: self-care, respiration and sphincter management, and mobility. The respiration and sphincter management subscale ranges from 0 to 40.
Function (mobility) as assessed by the Spinal Cord Independence Measure III Self Report (SCIM III SR) questionnaire | Pre-operative (5 repeated measurements over 2 months), post-operative at 2 weeks, 3 months, 6 months, 12 months, and 24 months
  The SCIM III SR is a measure of independence with activities across 3 subscales: self-care, respiration and sphincter management, and mobility. The mobility subscale ranges from 0 to 40.
Function as assessed total score on the Spinal Cord Independence Measure III Self Report (SCIM III SR) questionnaire | Pre-operative (5 repeated measurements over 2 months), post-operative at 2 weeks, 3 months, 6 months, 12 months, and 24 months
  The SCIM III SR is a measure of independence with activities across 3 subscales: self-care, respiration and sphincter management, and mobility. Total score ranges from 0 to 100( that is, the total score is the sum of scores on the three subscales).
Hand function as assessed by the Michigan Hand Questionnaire (MHQ) total score | Pre-operative, post-operative at 2 weeks, 3 months, 6 months, 12 months, and 24 months
  The MHQ instrument is a 37 core questions, self-report questionnaire used to assess changes in hand function. The MHQ requires subjects to rate their overall hand function, activities of daily living (ADLs), pain, work performance, aesthetics, and patient satisfaction with hand function. Scores on each of the 6 subscales range from 0 to 100, and an overall MHQ score is calculated by averaging the scores of the 6 subscales. The MHQ will be administered by the physicians or nurses involved in the study.
Hand function as assessed by the Sollerman Hand Function Test total score | Pre-operative, post-operative at 2 weeks, 3 months, 6 months, 12 months, and 24 months
  The Sollerman Hand Function Test is a standardized performance test designed to measure handgrips needed for certain activities of daily living (ADLs), such as eating, driving, personal hygiene, and writing. It includes multiple subtests that represent common handgrips and activities, completed using the hands both bilaterally and separately. Scoring of each subtest takes into account the time taken to complete the task, level of difficulty displayed, and quality of performance using correct grips. Scores range from 0 (task cannot be completed) - 4; a total score (0 - 80) is obtained from the sum of scores of all subtests.
Disability as assessed by the Disabilities of the Arm, Shoulder, and Hand (DASH) instrument total score | Pre-operative, post-operative at 2 weeks, 3 months, 6 months, 12 months, and 24 months
  The DASH instrument is a 30-item, self-report questionnaire used to assess overall upper extremity function. The DASH requires subjects to rate their ability to perform tasks using the upper extremities. Individuals are instructed to report their ability to perform the tasks, regardless of which arm they use or what strategies they employ. A single disability/symptom score is produced. Scores range from 0-100, where a greater score indicates greater disability. The DASH will be administered by the physicians, nurses, or physical therapist involved in the study.
Health-related Quality of Life as assessed by the Short Form 36 (SF-36) questionnaire total score | Pre-operative, post-operative at 2 weeks, 3 months, 6 months, 12 months, and 24 months
  The SF-36 is a questionnaire designed to measure general health and quality of life across eight, scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health)--a total score will be reported. The eight subscales are each given scores, which are the weighted sums of the questions in each subscale section, and each subscale score is directly transformed into a total score of 0-100 scale. The lower the score the more disability,a and the higher the score the less disability (that is, a score of zero is equivalent to maximum disability, and a score of 100 is equivalent to no disability). The SF-36 will be administered by the physicians, nurses, or physical therapist involved in the study.
Number of participants with intraoperative complications | 24 months
Number of participants with post-operative complications | 24 months
Number of participants who require reoperation | 24 months
Number of participants who receive the nerve transfer intervention soon after their spinal cord injury | at the time of the nerve transfer intervention
  The nerve transfer intervention will be considered "soon" or "early" if it is less than 12 months after the spinal cord injury that the nerve transfer intervention is intended to treat. This will be assessed at the time of the nerve transfer intervention.
Number of participants with an improvement in hand function as determined by qualitative video analysis | Pre-operative, post-operative at 6, 12, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Wesley H Jones, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States